CLINICAL TRIAL: NCT05884606
Title: A Prospective Pilot Study of the Allurion Digital Behaviour Change Intervention
Brief Title: The Allurion Digital Behaviour Change Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allurion Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRL-1000-0005
Record Dates: First submitted 2021-07-01; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Obesity
Keywords: Intragastric balloon
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Prospective Single Arm Cohort Pilot Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- non-randomized, pilot study (Experimental): This study is a prospective, non-randomized, pilot study to test the impact of the Allurion Digital Behaviour Change Intervention in participants who have been treated with the Allurion Gastric Balloon System. The study consists of the following segments:
  * Screening and enrolment period (prior to or day of Allurion Gastric Balloon System treatment)
  * All participants will take part in the Allurion DBCI for 6 months following study enrolment
  * All participants will complete a 6-month follow-up assessment after completion of the Allurion DBCI
  Interventions: Device: Allurion Digital Behaviour Change Intervention

INTERVENTIONS:
Device: Allurion Digital Behaviour Change Intervention — The Allurion DBCI adheres to current National Institute for Health and Care Excellence (NICE) guidance for obesity.

SUMMARY:
The proposed study is a prospective, non-randomized, pilot study to test the impact of the Allurion Digital Behaviour Change Intervention (DBCI) in participants who have been treated with the Allurion™ Gastric Balloon System. The study will include a nested qualitative and quantitative evaluations of the intervention from both the participant and Allurion provider perspective.

DETAILED DESCRIPTION:
The study consists of the following:

* Screening and enrolment period (prior to or day of Allurion Gastric Balloon System treatment)
* All participants will take part in the Allurion DBCI for 6 months following study enrolment
* All participants will complete a 6-month follow-up assessment after completion of the Allurion DBCI

ELIGIBILITY:
Inclusion Criteria:

* Allurion Gastric Balloon System placement in accordance with the approved Indications for Use
* Age 18 to 65 years of age
* BMI ≥ 27
* Weight < 180 kg
* Owns an Android or Apple smart phone
* Willing to download the Allurion App
* Willing to wear the Allurion Health Tracker Watch for the duration of the study
* Willing to use the Allurion Scale
* Proficient in reading the English language

Exclusion Criteria:

- Any condition contraindicated for the Allurion Gastric Balloon System as specified in the Instructions for Use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2021-06-19 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-11-06 (Actual)

PRIMARY OUTCOMES:
Change in percent total body weight loss (percent TBWL) | 6 months
  The primary outcome measure for this intervention is the change in percent total body weight loss (percent TBWL).

SECONDARY OUTCOMES:
Change in mental wellbeing | 6 and 12 months
  - Change in mental wellbeing as assessed by the The Warwick-Edinburgh Mental Well-being Scale. 14 (lowest mood) - 70 (highest mood)
Change in anxiety | 6 and 12 months
  - Change in anxiety as assessed by the the Generalized Anxiety Disorder scale. 0 (lowest anxiety) - 21 (highest anxiety)
Change in quality of life | 6 and 12 months
  - Change in quality of life as assessed by the Impact of Weight on Quality of Life-Lite Questionnaire Physical: 0 (lowest impact of weigh) - 28 (most impact of weight) Psychosocial: 0 (lowest impact of weight) - 52 (most impact of weight)
Change in loss of control over eating | 6 and 12 months
  - Change in loss of control over eating as assessed by the Loss of Control Over Eating Scale
  0 (most control of eating) - 28 (least control of eating)
Change in self-efficacy | 6 and 12 months
  - Change in self-efficacy as assessed by the Weight Efficacy Lifestyle Questionnaire 0 (least confidence in not overeating) - 80 (most confidence)
Change in barriers to exercise | 6 and 12 months
  - Change in barriers to exercise as assessed by the Barriers to Being Active Quiz 0 (least barriers to activity) - 12 (most barriers)
Time spent in physical activity steps (daily number of steps) | 6 and 12 months
  Time spent in physical activity will be measured by aerobic exercise (minutes) and steps (daily number of steps). This will be used in combination to assess physical activity.
Engagement with Health Coaching | 6 and 12 months
  Engagement with health coaching will be measured by categorization of the frequency and types of engagement interactions with participants. Categories of interactions will include both modes of delivery (e.g., messaging) and type of content (e.g., psychoeducation, behaviour change technique).
Engagement with the mobile and web app | 6 and 12 months
  Engagement with the mobile and web app will be measured by automated mobile and web App engagement will be measured by participant log-ins and number of chat messages with the health coach
Patient satisfaction | 6 and 12 months
  Patient self-reported intervention satisfaction via non-validated survey measures

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sacher, RD, PhD, Principal Investigator — Director
Locations (4):
- Netherlands (2):
  - Allurion Kliniek, Nederland, AB Hilversum
  - Nederlandse Obesitas Kliniek (NOK), Amsterdam
- United Kingdom (2):
  - Medizen Aesthetic Clinic, Sutton Coldfield, Birmingham
  - Monkhouse Surgical, Bromley, Kent

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers

REFERENCES:
- [Derived] Sacher PM, Fulton E, Rogers V, Wilson J, Gramatica M, Dent JE, Aarts EO, Eccleston D, Greve JW, Palm-Meinders I, Chuttani R. Impact of a Health Coach-Led, Text-Based Digital Behavior Change Intervention on Weight Loss and Psychological Well-Being in Patients Receiving a Procedureless Intragastric Balloon Program: Prospective Single-Arm Study. JMIR Form Res. 2024 Jul 31;8:e54723. doi: 10.2196/54723. PMID 39083340